CLINICAL TRIAL: NCT05173181
Title: Fixation of Displaced Distal Ulna Fractures in Adults by Flexible Intramedullary Nail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Hassan, Orthopedic Resident, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-11-08
Record Dates: First submitted 2021-11-27; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Fixation of Displaced Distal Ulna Fractures in Adults by Flexible Intramedullary Nail

STUDY DESIGN:
Intervention Model Description: The investigators have only one group of patients, (Adult with isolated fracture distal ulna). The investigators will do a single intervention, (Fixation with flexible intramedullary nail).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult with fracture distal ulna (Other)
  Interventions: Device: Flexible intramedullary nail

INTERVENTIONS:
Device: Flexible intramedullary nail — Fixation of distal ulna fracture with flexible intramedullary nail

SUMMARY:
The distal ulna is an important weight-bearing component of the wrist joint and an essential element of the forearm articulation. After injury, significant residual malalignment or deformity of the distal ulna and deficiency of its ligamentous support have a deleterious effect on grip strength and forearm rotation.

Although the best treatment option for displaced distal ulnar fracture remains a subject of debate, most surgeons aim for anatomical reduction and stable fixation to avoid disruption of the distal radioulnar joint.

The investigators will assess clinical and radiological results of fixation of displaced distal ulna fractures in adults by flexible intramedullary nail.

DETAILED DESCRIPTION:
The distal ulna is an important weight-bearing component of the wrist joint and an essential element of the forearm articulation. After injury, significant residual malalignment or deformity of the distal ulna and deficiency of its ligamentous support have a deleterious effect on grip strength and forearm rotation.

Fractures of the distal ulna usually occur in association with distal radius fractures.

Isolated distal ulnar fracture is an uncommon upper limb injury. It is usually the consequence of a direct blow against the soft tissue-deficient ulnar border.

Injuries to the distal ulna can lead to derangement of the distal radioulnar joint (DRUJ), subsequently resulting in pain from incongruity or ulnocarpal impaction, limitation of forearm rotation due to scarring, and weakness secondary to instability of the joint under load.

Isolated fractures of the distal third of the ulnar shaft can be treated successfully by conservative if not significantly displaced and if rotational malalignment is not present. Fractures with significant displacement or those with rotational malalignment (displaced spiral fracture patterns) are best be treated by osteosynthesis and functional rehabilitation in order to prevent loss of forearm rotation.

Although the best treatment option for displaced distal ulnar fracture remains a subject of debate, most surgeons aim for anatomical reduction and stable fixation to avoid disruption of the distal radioulnar joint.

The investigators aim is to assess clinical and radiological results of fixation of displaced distal ulna fractures in adults by flexible intramedullary nail.

It is a prospective study patients with displaced distal ulna fractures in adult patient admitted in orthopaedic department of Sohag University Hospital after taking an informed consent from patients or near relatives. Fractures will be managed using flexible intra medullary nail .

Patients with Intra articular fractures , Fractures with disturbed radioulnar joint , or Old malunited or deformed distal ulna are excluded.

* Clinical evaluation of patient by Grace and Eversmann rating system used to assess functional evaluation ,VAS (visual analogue scale),or Dash score (Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire scores).
* Radiological evaluation as plain x ray.

Time plan : clinical and radiolodical evaluation as follow:

* Immediately postoperative.
* 2 weeks postoperative.
* 1month postoperative.
* 2 months postoperative.
* 6 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Patients with displaced distal ulna fractures in adult patient admitted in orthopaedic department of Sohag University Hospital after taking an informed consent from patients or near relatives

Exclusion Criteria:

* Patients with Intra articular fractures
* Fractures with disturbed radioulnar joint
* Old malunited or deformed distal ulna

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Radiological evaluation | Immediately postoperative
  Displacement of fracture - signs of healing
Grace and Eversmann rating system | 6 months postoperative
  Rating system that was based only on fracture union and pronation-supination of the forearm. Motion of the wrist and elbow was not used in the rating system, 10 means excellent results 4 means acceptable results.
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire scores | 6 months postoperative
  Self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100
Radiological evaluation | 2 weeks postoperative
  Displacement of fracture - signs of healing
Radiological evaluation | 1month postoperative
  Displacement of fracture - signs of healing
Radiological evaluation | 2 months postoperative
  Displacement of fracture - signs of healing
Radiological evaluation | 6 months postoperative
  Displacement of fracture - signs of healing

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet

REFERENCES:
- [Result] Grace TG, Eversmann WW Jr. Forearm fractures: treatment by rigid fixation with early motion. J Bone Joint Surg Am. 1980 Apr;62(3):433-8. PMID 7364814
- [Result] Matthews LS, Kaufer H, Garver DF, Sonstegard DA. The effect on supination-pronation of angular malalignment of fractures of both bones of the forearm. J Bone Joint Surg Am. 1982 Jan;64(1):14-7. PMID 7054197
- [Result] PATRICK J. A study of supination and pronation, with especial reference to the treatment of forearm fractures. J Bone Joint Surg Am. 1946 Oct;28(4):737-48. No abstract available. PMID 21003183